CLINICAL TRIAL: NCT01289769
Title: The Effect of Prophylactic Dexmedetomidine on Hemodynamic Disturbances During Double Lumen Endotracheal Intubation. A Double-blinded, Randomized, Placebo-Controlled Trial.
Brief Title: The Effect of Dexmedetomidine on Hemodynamic Response During Double Lumen Endotracheal Intubation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Tanyong Pipanmekaporn, Department of Anesthesiology, Faculty of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COM-10-11-19B-11; research ID 77 (Other: Research ID 77)
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Intubation Complication; Tracheal Intubation Morbidity; Anesthesia Intubation Complication; Hypertension; High Blood Pressure; Tachycardia
MeSH Terms: conditions — Hypertension; Tachycardia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine 0.7 microgram per kilogram in saline 20 ml given within 10 minutes before intubation
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: Placebo — normal saline 20 ml( the same volume as dexmedetomidine) giving within 10 minutes.
  Arms: control

SUMMARY:
The purpose of this study is to evaluate the effect of dexmedetomidine on hemodynamic responses during laryngoscopy and double lumen endotracheal intubation and assess the adverse effect related to complications of dexmedetomidine.

DETAILED DESCRIPTION:
The cardiovascular responses to laryngoscopy and tracheal intubation are mediated by both sympathetic and parasympathetic nervous system. The hemodynamic responses resulting from sympathetic nervous system stimulation are tachycardia, cardiac arrhythmias, hypertension, increased intraocular pressure, increased intracranial pressure, bronchospasm and myocardial ischemia. Tachycardia is one of the major predictor of intraoperative myocardial ischemia and causes an imbalance of myocardial oxygen supply and demand. Although hemodynamic responses to laryngoscopy and intubation is transient, these effect may be harmful to patients suffering from myocardial and cerebrovascular diseases. The placement of double lumen endotracheal tube may produce similar or greater pressor response than endotracheal tube because of larger sizes and greater carinal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status I-III
* Undergoing Elective Thoracotomy or Thoracoscopy
* Required Left Sided-double Lumen Endotracheal Intubation

Exclusion Criteria:

* Patients with bradycardia (heart rate < 50 beat per minute) or heart block
* Suspected of Difficult Intubation
* Patients Who Are at Risk for Rapid Change of Hemodynamics
* Allergic to Dexmedetomidine
* Hepatic or Renal Impairment (Preoperative Serum Creatinine > 1.5 mg/dl)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change in systolic blood pressure | (day 1) before induction, before intubation and every minute for the first 10 minutes after endotracheal intubation
  direct arterial pressure monitoring
change in diastolic blood pressure | (day 1) before induction, before intubation and every minute for the first 10 minutes after endotracheal intubation
  direct arterial pressure monitoring
change in mean arterial pressure | (day 1) before induction, before intubation and every minute for the first 10 minutes after endotracheal intubation
  direct arterial pressure monitoring
change in heart rate | (day 1) before induction, before intubation and every minute for the first 10 minutes after endotracheal intubation

SECONDARY OUTCOMES:
adverse events related to dexmedetomidine | (day 1) during dexmedetomidine administration until 10 minutes after endotracheal intubation
  bradycardia, hypotension, arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Tanyong Pipanmekaporn, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Chiang Mai University , Chiang Mai, Thailand,50200
Locations (1):
- Chiang Mai University Hospital, Maung, Chiang Mai, Thailand

REFERENCES:
- [Background] Basar H, Akpinar S, Doganci N, Buyukkocak U, Kaymak C, Sert O, Apan A. The effects of preanesthetic, single-dose dexmedetomidine on induction, hemodynamic, and cardiovascular parameters. J Clin Anesth. 2008 Sep;20(6):431-6. doi: 10.1016/j.jclinane.2008.04.007. PMID 18929283
- [Background] Maguire A, Thompson JP, Guest C, Sadler PJ, Strupish JW, West KJ. Comparison of the effects of intravenous alfentanil and esmolol on the cardiovascular response to double-lumen endobronchial intubation. Anaesthesia. 2001 Apr;56(4):319-25. doi: 10.1046/j.1365-2044.2001.01917.x. PMID 11284817
- [Derived] Pipanmekaporn T, Punjasawadwong Y, Charuluxananan S, Lapisatepun W, Bunburaphong P. The effect of prophylactic dexmedetomidine on hemodynamic disturbances to double-lumen endotracheal intubation: a prospective, randomized, double-blind, and placebo-controlled trial. Anesthesiol Res Pract. 2013;2013:236089. doi: 10.1155/2013/236089. Epub 2013 Jul 29. PMID 23983684